CLINICAL TRIAL: NCT00244751
Title: A Double-Blind, Randomized, Placebo-Controlled Multi-Center, Phase II Parallel Dose-Ranging Study to Assess the Antifibrotic Activity of GI262570 in Chronic Hepatitis C Subjects With Hepatic Fibrosis Who Have Failed Prior Antiviral Therapy
Brief Title: Antifibrotic Activity Of GI262570 In Chronic Hepatitis C Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: FBX104114
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Cirrhosis, Liver
Keywords: Hepatitis C liver fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — farglitazar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GI262570 0.5 mg (Experimental): Participants received GI262570 0.5 milligrams (mg) tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
  Interventions: Drug: GI262570 0.5 mg
- GI262570 1.0 mg (Experimental): Participants received GI262570 1.0 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
  Interventions: Drug: GI262570 1.0 mg
- Placebo (Placebo Comparator): Participants received matching placebo tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GI262570 0.5 mg — GI262570 0.5 mg
  Arms: GI262570 0.5 mg
Drug: GI262570 1.0 mg — GI262570 1.0 mg
  Arms: GI262570 1.0 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety and effectiveness of GI262570 compared to placebo (a pill that looks exactly like GI262570 but contains no active medicine) in improving specific tests that indicate the degree of liver fibrosis (scarring). Subjects who are enrolled in the study must have had prior treatment with interferon (either pegylated or standard interferon) plus ribavirin for at least 12 weeks to treat their hepatitis C, but either failed to clear the virus or didn't tolerate the treatment.

ELIGIBILITY:
Inclusion criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Age between 40 and 70 years, inclusive.
* Documented positive serology for HCV antibody by a second generation or higher assay.
* Serum HCV RNA positive and HCV viral Genotype 1 at pre-screening visit.
* Ishak fibrosis score of 2, 3 or 4.
* Failure to achieve sustained virologic response (SVR) with previous interferon (standard or pegylated) and ribavirin treatment administered at a minimum dose of 3mU three times weekly or equivalent, for at least 12 weeks. Reasons for failure may include failure to respond to treatment or intolerability to optimal treatment. Prior treatment with interferon/ribavirin must have been discontinued at least 11 months prior to the biopsy date.
* Male or female; a female is eligible to enter and participate in this study if she is of:

  1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
  2. child-bearing potential, has a negative serum pregnancy test at screen, and agrees to one of the following:

     * Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the investigational drug, (a minimum of 5 half-lives or longer if the pharmacodynamic profile of the investigational drug warrants a longer time period); or,
     * Female sterilization; or,
     * Has a male partner who is sterilized; or,
     * Implants of levonorgestrel; or,
     * Injectable progestogen; or,
     * Oral contraceptive (combined or progestogen only) , must be stable for 3 months prior to study entry; or,
     * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or,
     * Any other methods with published data showing that the lowest expected failure rate for that method is less than 1% per year; or,
     * Barrier method only if used in combination with any of the above acceptable methods.
* Availability and willingness of subject to provide written informed consent.

Exclusion criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* History of ascites, variceal hemorrhage, hepatic encephalopathy, spontaneous bacterial peritonitis or other signs of hepatic decompensation.
* Current or historical evidence suggestive of ischemic heart disease or other cardiovascular disease that in the investigator's opinion may adversely impact the safety of the subject during the conduct of the study. Evidence suggestive of cardiovascular disease may come from a number of sources, including clinical history, physical exam, electrocardiogram, laboratory testing, and radiographic procedures.
* New York Heart Association (NYHA) Functional Class 1, 2, 3, or 4 cardiac status
* Co-infection with HBV or HIV.
* Liver histology consistent with any other co-existing cause of chronic liver disease.
* Documented evidence of a hepatic mass lesion suspicious for hepatocellular carcinoma.
* Alpha-fetoprotein > 200ng/mL at pre-screening.
* Inadequate hematologic function defined by any of the following:

Hemoglobin (<12.5 g/dL for men)(<12.0 g/dL for women)

Absolute Neutrophil Count (ANC) (<1.0 x 10^9/L) Platelets (<130X/10^9/L)

* Inadequate renal function defined as:

Serum creatinine (>1.5mg/dL (≥130mmol/L)) Calculated creatinine clearance as calculated by Cockcroft and Gault (<60mL/min)

* Serum ALT level ≥5 x ULN.
* Albumin <3.2g/dL.
* Total bilirubin >1.2 x ULN.
* Prothrombin time > 15 seconds or International normalized ratio (INR) > 1.3.
* Organ, stem cell, or bone marrow transplant.
* Serious concurrent medical illness that in the investigator's opinion might interfere with therapy. This includes significant systemic illnesses (other than liver disease) such as chronic pancreatitis.
* Active systemic autoimmune disorder.
* A pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or renal function that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* Other medical conditions that, in the investigator's opinion, might interfere with compliance with therapy, participation in the study or interpretation of results.
* Pregnancy (or lactation) or, in subjects capable of bearing children, inability/unwillingness to practice adequate contraception.
* Females of child-bearing potential (post-puberty) unwilling or unable to have pregnancy testing at any study visit.
* Therapy with systemic cytotoxic agents, immunomodulators, or immunosuppressive therapy requiring use of more than 5mg of prednisone (or its equivalent) per day.
* Therapy with a systemic antiviral agent (with the exception of prophylaxis or treatment of influenza or chronic HSV) within the past 30 days.
* Concurrent participation in another clinical trial in which the subject is or will be exposed to another investigational or a non-investigational drug or device within 30 days of the screening visit.
* Current therapy or anticipated need for therapy with hypoglycemic drugs (e.g., insulin, sulfonylurea or metformin).
* Known hypersensitivity to GI262570, or to any component of the GI262570 soft gelatin capsules, dispersion tablets or the sodium salt tablet or to PPARg agonists.
* A history of hepatotoxicity to TZDs and/or a history of severe edema or medically serious fluid-related events associated with the use of TZDs.
* Use of other PPAR agonists (e.g., rosiglitazone, pioglitazone) within 1 year from the start of dosing.
* Active alcohol abuse within the past 1 year.
* Use of illegal drugs in the past 1 year. 30a. Macular edema or history of macular edema.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2005-11-02 (Actual); Primary Completion 2008-03-13 (Actual); Study Completion 2008-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (101):
- United States (48):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, North Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Clemente, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Lutherville-Timonium, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Australia (6):
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Camperdown, Victoria
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Fitzroy, Melbourne, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Canada (9):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Czechia (3):
  - GSK Investigational Site, Brno-Bohunice
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Prague
- Germany (14):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Israel (6):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Nazareth
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Malaysia (2):
  - GSK Investigational Site, Bandar Tun Razak, Cheras
  - GSK Investigational Site, Kepong
- GSK Investigational Site, Auckland, New Zealand
- GSK Investigational Site, San Juan, Puerto Rico
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca, Cluj
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Singapore, Singapore
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in North America, Europe, and the International region. There were 22 study sites in Europe, 9 study sites in the International region and 45 study sites in North America. The study was conducted duration 02-November-2005 to 03-March-2008.
Pre-assignment Details: The study consisted of a pre-screening visit (within 60 days of first dose) and a screen visit. For this study, 110 sites screened 863 participants. Of these participants, 265 were randomized.
Period: Overall Study
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Started | 88 | 89 | 88
Completed | 72 | 74 | 78
Not Completed | 16 | 15 | 10
Not completed — Adverse Event | 7 | 7 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 5 | 3
Not completed — Elevated liver enzymes | 1 | 0 | 0
Not completed — Lack of compliance with protocol | 0 | 1 | 0
Not completed — Safety reasons | 0 | 1 | 0
Not completed — Participant randomized by mistake | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GI262570 0.5 mg: Participants received GI262570 0.5 mg. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
- GI262570 1.0 mg: Participants received GI262570 1.0 mg once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
- Total: Total of all reporting groups
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg | Total
Number analyzed (Participants) | 88 | 89 | 88 | 265
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (5.64) | 52.2 (7.25) | 51.4 (5.81) | 51.9 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 29 | 100
  Male | 53 | 53 | 59 | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 3 | 7
  Asian | 11 | 6 | 7 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 14 | 9 | 35
  White | 63 | 67 | 68 | 198
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Liver Biopsy Immunohistochemical Marker of Hepatic Stellate Cell (HSC) Activation and Collagen Synthesis at Week 52
Description: A percutaneous liver biopsy was obtained at the screening visit and at Week 52. A new liver biopsy at the screening visit was not taken in the event that a previous liver biopsy taken within 120 days of the Baseline /Day 1 visit (day of first dose), and the tissue block was available. The immunohistochemical marker assessed was smooth muscle alpha-actin (aSMA). Sections of the liver biopsies were stained by standard immunocytochemical techniques using a monoclonal antibody to smooth muscle actin with 'very intense purple' as the detection chromogen. This gives a reddish-purple color to the activated stellate cells, which strongly contrasts with the rest of the tissue. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing. The values are presented as proportion of positive area over total area.
Time Frame: Baseline and Week 52
Population: Modified Intent to Treat (MITT) Population consisted of all participants with chronic hepatitis C randomized, regardless of whether or not the study drug was actually taken or if the participant completed the planned duration of the study. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio of positive area
Groups:
- GI262570 0.5mg: Participants received GI262570 0.5 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
- GI262570 1.0mg: Participants received GI262570 1.0 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
Arm/Group | Placebo | GI262570 0.5mg | GI262570 1.0mg
Number analyzed (Participants) | 64 | 71 | 72
Ratio of positive area | 0.02065 (0.047620) | 0.02819 (0.048160) | 0.02914 (0.040948)
Statistical Analysis 1: Comparison: Placebo vs GI262570 0.5mg; Test type: Superiority or Other; p = 0.3608, reduced regression model
Statistical Analysis 2: Comparison: Placebo vs GI262570 1.0mg; Test type: Superiority or Other; p = 0.3575, reduced regression model

2. Primary Outcome: Mean Change From Baseline in Fibrosis as Quantified by Morphometric Image Analysis
Description: A percutaneous liver biopsy was obtained at the screening visit and at Week 52. A new liver biopsy at the screening visit was not taken in the event that a previous liver biopsy taken within 120 days of the Baseline /Day 1 visit (day of first dose), and the tissue block was available. Morphometric analysis was performed using specimens stained with Sirius red and computerized image analysis. Sirius red was used to stain extracellular collagen in liver sections. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing. The values are presented as proportion of positive area over total area.
Time Frame: Baseline and at Week 52
Population: MITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio of positive area
Groups:
- GI262570 0.5 mg: Participants received GI262570 0.5 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 65 | 71 | 72
Ratio of positive area | 0.02541 (0.058338) | 0.02613 (0.055985) | 0.02527 (0.060665)
Statistical Analysis 1: Comparison: Placebo vs GI262570 0.5 mg; Test type: Superiority or Other; p = 0.9157, reduced regression model
Statistical Analysis 2: Comparison: Placebo vs GI262570 1.0 mg; Test type: Superiority or Other; p = 0.9501, reduced regression model

3. Primary Outcome: Number of Participants With Ranked Histological Assessment of the Paired Biopsies at Week 52
Description: In ranked assessment (fibrosis and necroinflammation), available slides from each participant were evaluated as to whether one slide presents a globally more benign histopathology or whether the matched slides comprise globally equivalent histologic patterns. Subsequent data analysis revealed whether slides scored (within matched pairs of slides) as more benign occurred in different proportions of the Week 52 liver biopsies, according to treatment group. The number of participants with paired biopsies was based on the number with a Rank Assessment.
Time Frame: Week 52
Population: MITT Population. Only those participants with paired biopsies at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GI262570 0.5mg | GI262570 1.0mg
Number analyzed (Participants) | 65 | 72 | 72
Participants
  Fibrosis, better than screening | 13 | 17 | 11
  Fibrosis, same as screening | 35 | 38 | 35
  Fibrosis, worse than screening | 16 | 17 | 25
  Fibrosis, missing | 1 | 0 | 1
  Necrosis, better than screening | 11 | 20 | 27
  Necrosis, same as screening | 23 | 24 | 23
  Necrosis, worse than screening | 31 | 28 | 22
  Necrosis, missing | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs GI262570 0.5mg vs GI262570 1.0mg; Comparison for Ranked assessment (fibrosis); Test type: Superiority or Other; p = 0.6483, Cochran-Mantel-Haenszel Test
Statistical Analysis 2: Comparison: Placebo vs GI262570 0.5mg vs GI262570 1.0mg; Comparison for Ranked assessment (necrosis); Test type: Superiority or Other; p = 0.1776, Cochran-Mantel-Haenszel Test

4. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to 4 weeks post treatment (52 weeks)
Population: As Treated Population consisted of all participants for whom no clear evidence was available of failure to take study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GI262570 0.5mg | GI262570 1.0mg
Number analyzed (Participants) | 88 | 89 | 88
Participants
  Any AE | 75 | 68 | 71
  Any SAE | 7 | 10 | 6

5. Primary Outcome: Number of Participants With Abnormal ECG Findings
Description: A standardized 12-lead ECGs were recorded at pre-screening, and pre-dose, at Baseline/Day 1, Weeks 16, 34, and 52 or withdrawal and at the 4 week follow-up visit. Any conditions such as bundle branch block, repolarization, depolarization, abnormal sinus rhythms, atrial fibrillation etc. are considered to be clinically abnormal findings.
Time Frame: Up to 4 weeks post-treatment (52 weeks)
Population: As Treated Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GI262570 0.5mg | GI262570 1.0mg
Number analyzed (Participants) | 88 | 89 | 88
Participants
  Baseline, Abnormal, not clinically significant: number analyzed (Participants) | 86 | 88 | 87
  Baseline, Abnormal, not clinically significant | 25 | 25 | 22
  Week 16, Abnormal, not clinically significant: number analyzed (Participants) | 76 | 82 | 83
  Week 16, Abnormal, not clinically significant | 18 | 16 | 21
  Week 34, Abnormal, not clinically significant: number analyzed (Participants) | 72 | 77 | 78
  Week 34, Abnormal, not clinically significant | 12 | 19 | 23
  Week 34, Abnormal, clinically significant: number analyzed (Participants) | 72 | 77 | 78
  Week 34, Abnormal, clinically significant | 0 | 0 | 1
  Week 52, Abnormal, not clinically significant: number analyzed (Participants) | 71 | 75 | 75
  Week 52, Abnormal, not clinically significant | 10 | 18 | 22

6. Primary Outcome: Number of Participants With Change in Toxicities Grades 3 and 4 of Laboratory Parameters Over Time
Description: Clinical laboratory parameters: Alkaline phosphatase, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Total bilirubin, Cholesterol, Carbon dioxide content/Bicarbonate (CO2/HCO3), Creatinine, Glucose, Hemoglobin, Potassium, Low density lipid (LDL) cholesterol, Lymphocytes, Sodium, Segmented neutrophils, Platelet count, White blood cell (WBC) count were assessed for change in grade toxicities. Toxicities were graded as grade 1 to grade 4 in increasing order of severity of toxicity. Thus grade 4 indicating severe toxicity. Only those parameters with grade 3 and 4 toxicities are presented.
Time Frame: Up to 4 weeks post-treatment (52 weeks)
Population: As Treated Population. Only those participants available at the specified time points for particular parameter were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 88 | 89 | 88
Participants
  ALT, grade 3: number analyzed (Participants) | 55 | 56 | 58
  ALT, grade 3 | 4 | 2 | 5
  ALT, grade 4: number analyzed (Participants) | 55 | 56 | 58
  ALT, grade 4 | 1 | 0 | 0
  AST, grade 3: number analyzed (Participants) | 56 | 61 | 52
  AST, grade 3 | 4 | 2 | 2
  AST, grade 4: number analyzed (Participants) | 56 | 61 | 52
  AST, grade 4 | 1 | 0 | 0
  Total bilirubin, grade 4: number analyzed (Participants) | 16 | 19 | 25
  Total bilirubin, grade 4 | 12 | 17 | 22
  Glucose, grade 3: number analyzed (Participants) | 87 | 89 | 86
  Glucose, grade 3 | 1 | 0 | 0
  Glucose, grade 4: number analyzed (Participants) | 87 | 89 | 86
  Glucose, grade 4 | 0 | 1 | 0
  Hemaglobin, grade 3: number analyzed (Participants) | 0 | 3 | 3
  Hemaglobin, grade 3 |  | 1 | 1
  Potassium, grade 4: number analyzed (Participants) | 87 | 89 | 86
  Potassium, grade 4 | 1 | 0 | 0
  Sodium, grade 4: number analyzed (Participants) | 87 | 89 | 86
  Sodium, grade 4 | 1 | 1 | 1
  Segmented neutrophils, grade 4: number analyzed (Participants) | 7 | 4 | 3
  Segmented neutrophils, grade 4 | 1 | 0 | 0
  Platelet count, grade 4: number analyzed (Participants) | 11 | 6 | 11
  Platelet count, grade 4 | 1 | 0 | 0

7. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DSP)
Description: SBP and DBP readings were taken at pre-screening, pre-dose after 10 minutes of rest, at Baseline/Day 1, weeks 2, 4, 10, 16, 22, 28, 34, 40, 46, and 52 or WD and at the 4 week follow-up visit. Day 1 (before dosing) value was considered to be as Baseline value. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing.
Time Frame: Baseline and up to 4 weeks post-treatment (52 weeks)
Population: As Treated Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 88 | 89 | 88
Millimeter of mercury
  DBP, Week 2: number analyzed (Participants) | 86 | 85 | 86
  DBP, Week 2 | -0.06 (12.347) | 0.60 (9.129) | 0.17 (8.171)
  DBP, Week 4: number analyzed (Participants) | 85 | 87 | 85
  DBP, Week 4 | 1.12 (8.793) | -1.31 (7.560) | -0.02 (8.018)
  DBP, Week 10: number analyzed (Participants) | 83 | 86 | 84
  DBP, Week 10 | 0.94 (9.195) | -1.62 (10.032) | 0.00 (7.309)
  DBP, Week 16: number analyzed (Participants) | 78 | 84 | 83
  DBP, Week 16 | 0.31 (9.194) | -2.00 (9.664) | 0.06 (8.226)
  DBP, Week 22: number analyzed (Participants) | 78 | 81 | 81
  DBP, Week 22 | 1.18 (10.264) | -2.46 (9.648) | 0.93 (8.194)
  DBP, Week 28: number analyzed (Participants) | 76 | 79 | 81
  DBP, Week 28 | 0.87 (10.529) | -1.09 (9.664) | 0.15 (9.231)
  DBP, Week 34: number analyzed (Participants) | 75 | 77 | 79
  DBP, Week 34 | 0.40 (11.480) | -1.38 (9.242) | 0.70 (8.612)
  DBP, Week 40: number analyzed (Participants) | 74 | 76 | 79
  DBP, Week 40 | 0.05 (10.136) | -2.20 (8.947) | 1.16 (9.302)
  DBP, Week 46: number analyzed (Participants) | 74 | 73 | 79
  DBP, Week 46 | 0.95 (10.620) | -1.16 (9.203) | 1.29 (8.423)
  DBP, Week 52: number analyzed (Participants) | 72 | 74 | 76
  DBP, Week 52 | -0.01 (10.177) | -0.64 (9.807) | -0.13 (6.855)
  DBP, Withdrawal: number analyzed (Participants) | 11 | 9 | 6
  DBP, Withdrawal | 2.45 (9.015) | 0.89 (8.852) | 1.00 (5.933)
  DBP, post-treatment: number analyzed (Participants) | 80 | 77 | 82
  DBP, post-treatment | 0.66 (11.085) | -0.29 (10.860) | 0.49 (9.634)
  SBP, Week 2: number analyzed (Participants) | 86 | 85 | 86
  SBP, Week 2 | 0.17 (16.700) | -0.53 (14.095) | 0.49 (12.516)
  SBP, Week 4: number analyzed (Participants) | 85 | 87 | 85
  SBP, Week 4 | 0.78 (16.821) | -1.34 (13.333) | -0.80 (12.343)
  SBP, Week 10: number analyzed (Participants) | 83 | 86 | 84
  SBP, Week 10 | 2.95 (16.888) | -0.47 (14.524) | -0.85 (13.293)
  SBP, Week 16: number analyzed (Participants) | 78 | 84 | 83
  SBP, Week 16 | 0.83 (15.621) | -1.79 (15.496) | 0.10 (11.008)
  SBP, Week 22: number analyzed (Participants) | 78 | 81 | 81
  SBP, Week 22 | 0.45 (18.161) | -1.79 (14.361) | 0.59 (12.217)
  SBP, Week 28: number analyzed (Participants) | 76 | 79 | 81
  SBP, Week 28 | -1.82 (20.285) | -2.16 (15.260) | 1.69 (14.782)
  SBP, Week 34: number analyzed (Participants) | 75 | 77 | 79
  SBP, Week 34 | 0.95 (19.558) | -1.86 (15.059) | 0.32 (13.569)
  SBP, Week 40: number analyzed (Participants) | 74 | 76 | 79
  SBP, Week 40 | -1.34 (19.616) | -1.04 (13.085) | -1.23 (14.371)
  SBP, Week 46: number analyzed (Participants) | 74 | 73 | 79
  SBP, Week 46 | -0.53 (15.173) | -1.85 (12.158) | 0.30 (13.670)
  SBP, Week 52: number analyzed (Participants) | 72 | 74 | 76
  SBP, Week 52 | 0.15 (18.950) | 1.92 (13.352) | -0.21 (12.414)
  SBP, Withdrawal: number analyzed (Participants) | 11 | 9 | 6
  SBP, Withdrawal | 5.09 (25.126) | -0.44 (21.830) | -0.17 (3.488)
  SBP, Post-treatment: number analyzed (Participants) | 80 | 77 | 82
  SBP, Post-treatment | 0.25 (21.747) | 1.69 (13.431) | 3.52 (16.931)

8. Primary Outcome: Mean Change From Baseline in Heart Rate
Description: Heart rate assessment were done at pre-screening, pre-dose after 10 minutes of rest, at Baseline/Day 1, weeks 2, 4, 10, 16, 22, 28, 34, 40, 46, and 52 or WD and at the 4 week follow-up visit. Day 1 (before dosing) value was considered to be as Baseline value. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to be missing.
Time Frame: Baseline and up to 4 weeks post-treatment (52 weeks)
Population: As treated population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 88 | 89 | 88
beats per minute
  Week 2: number analyzed (Participants) | 86 | 85 | 86
  Week 2 | 1.08 (8.763) | -1.92 (7.143) | -0.28 (8.554)
  Week 4: number analyzed (Participants) | 85 | 87 | 85
  Week 4 | 0.35 (9.726) | 0.55 (10.223) | 1.80 (10.221)
  Week 10: number analyzed (Participants) | 83 | 86 | 84
  Week 10 | 2.04 (8.824) | 0.49 (8.771) | 0.83 (8.747)
  Week 16: number analyzed (Participants) | 78 | 84 | 83
  Week 16 | -0.44 (8.425) | -0.33 (9.295) | 0.55 (11.070)
  Week 22: number analyzed (Participants) | 78 | 81 | 81
  Week 22 | 2.23 (9.120) | -0.10 (10.706) | 3.23 (12.141)
  Week 28: number analyzed (Participants) | 76 | 79 | 81
  Week 28 | 0.80 (8.857) | -1.54 (8.530) | 0.05 (8.237)
  Week 34: number analyzed (Participants) | 75 | 77 | 79
  Week 34 | 0.89 (9.983) | 0.77 (9.485) | -0.13 (10.655)
  Week 40: number analyzed (Participants) | 74 | 76 | 78
  Week 40 | -0.11 (8.340) | -1.89 (9.169) | 0.09 (11.101)
  Week 46: number analyzed (Participants) | 74 | 73 | 79
  Week 46 | 1.18 (9.411) | -1.01 (10.360) | 1.08 (12.056)
  Week 52: number analyzed (Participants) | 72 | 74 | 76
  Week 52 | 1.04 (9.300) | -0.26 (9.656) | -2.09 (12.197)
  Withdrawal: number analyzed (Participants) | 11 | 9 | 6
  Withdrawal | 5.27 (14.107) | 1.00 (12.062) | -1.17 (3.061)
  Post-treatment: number analyzed (Participants) | 80 | 77 | 82
  Post-treatment | 1.20 (10.184) | -0.42 (10.287) | 0.15 (11.340)

9. Primary Outcome: Number of Participants With Fluid Retention Events
Description: Fluid retention event was one of the AEs reported. AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 4 weeks post-treatment (52 weeks)
Population: As Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GI262570 0.5mg | GI262570 1.0mg
Number analyzed (Participants) | 88 | 89 | 88
Participants | 0 | 1 | 1

10. Secondary Outcome: Number of Participants Progressing at Least 1 Point on the Ishak Fibrosis Score at Week 52
Description: Progression was defined as an increase by at least one point in the fibrosis score. Score ranged from 0 to 6 (higher score indicates greater fibrosis). 0: No fibrosis, 1: Fibrous expansion of some portal areas, with or without short fibrous septa, 2: Fibrous expansion of most portal areas, with or without short fibrous septa, 3: Fibrous expansion of most portal areas with portal to portal bridging, 4: Fibrous expansion of portal areas with marked bridging, 5: Marked bridging with occasional nodules (incomplete cirrhosis), 6: Cirrhosis, probable or definite. The number of participants with paired biopsies is based on the number with an Ishak Fibrosis score.
Time Frame: Week 52
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Groups:
- GI262570 1.0mg: Participants received GI262570 1.0 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.Participants received GI262570 1.0 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
Arm/Group | Placebo | GI262570 0.5mg | GI262570 1.0mg
Number analyzed (Participants) | 64 | 72 | 71
Participants | 12 | 14 | 19

11. Secondary Outcome: Number of Participants Regressing at Least 1 Point on the Ishak Fibrosis Score at Week 52
Description: Regression was defined as a decrease by at least one point in the fibrosis score. Score ranged from 0 to 6 (higher score indicates greater fibrosis). 0: No fibrosis, 1: Fibrous expansion of some portal areas, with or without short fibrous septa, 2: Fibrous expansion of most portal areas, with or without short fibrous septa, 3: Fibrous expansion of most portal areas with portal to portal bridging, 4: Fibrous expansion of portal areas with marked bridging, 5: Marked bridging with occasional nodules (incomplete cirrhosis), 6: Cirrhosis, probable or definite. The number of participants with paired biopsies is based on the number with an Ishak Fibrosis score.
Time Frame: Week 52
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 64 | 72 | 71
Participants | 11 | 14 | 9

12. Secondary Outcome: Number of Participants Whose Ishak Fibrosis Score Remains Unchanged at Week 52
Description: No change was defined as having the same score at both Baseline and at Week 52. Score ranged from 0 to 6 (higher score indicates greater fibrosis). 0: No fibrosis, 1: Fibrous expansion of some portal areas, with or without short fibrous septa, 2: Fibrous expansion of most portal areas, with or without short fibrous septa, 3: Fibrous expansion of most portal areas with portal to portal bridging, 4: Fibrous expansion of portal areas with marked bridging, 5: Marked bridging with occasional nodules (incomplete cirrhosis), 6: Cirrhosis, probable or definite. The number of participants with paired biopsies is based on the number with an Ishak Fibrosis score.
Time Frame: Week 52
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 64 | 72 | 71
Participants | 41 | 44 | 43

13. Secondary Outcome: Mean Change From Screening in Total Ishak Score (Necroinflammatory Score and Fibrosis Score) at Week 52
Description: Ishak score ranged from 0 to 6 (higher score indicates greater fibrosis). 0: No fibrosis, 1: Fibrous expansion of some portal areas, with or without short fibrous septa, 2: Fibrous expansion of most portal areas, with or without short fibrous septa, 3: Fibrous expansion of most portal areas with portal to portal bridging, 4: Fibrous expansion of portal areas with marked bridging, 5: Marked bridging with occasional nodules (incomplete cirrhosis), 6: Cirrhosis, probable or definite. The necroinflammatory score is the combined score for necrosis and inflammation domains and ranged from 0 (best) to 14 (worst). Change from screening was calculated as the post screening assessment minus the screening assessment for a given parameter.
Time Frame: Screening and Week 52
Population: MITT Population. Only those participants available at the specified time point were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 88 | 89 | 88
Scores on a scale
  Necroinflammatory Score: number analyzed (Participants) | 65 | 72 | 72
  Necroinflammatory Score | 0.7 (1.31) | 0.2 (1.60) | -0.2 (1.69)
  Fibrosis Score: number analyzed (Participants) | 64 | 72 | 71
  Fibrosis Score | 0.1 (0.71) | 0.0 (0.85) | 0.2 (0.70)

14. Secondary Outcome: Mean Change From Screening in Metavir Scores at Week 52
Description: Metavir activity score ranged from 0 to 3 (higher score indicates severe symptoms of necrosis). 0: Piecemeal necrosis (PMN) absent and lobular necrosis (LN) absent or slight, 1: PMN slight and LN moderate, 2: PMN moderate and LN severe, 3: PMN severe. Metavir fibrosis score ranged from 0 to 4 (higher score indicates severe symptoms of necrosis). 0: No fibrosis, 1: Portal fibrosis without septa, 2: Portal fibrosis with septa, 3: Septal fibrosis without cirrhosis, 4: Cirrhosis. Change from screening was calculated as the post screening assessment minus the screening assessment for a given parameter.
Time Frame: Screening and Week 52
Population: MITT Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 88 | 89 | 88
Scores on a scale
  Metavir: Activity: number analyzed (Participants) | 65 | 72 | 72
  Metavir: Activity | 0.18 (0.556) | -0.01 (0.722) | -0.04 (0.680)
  Metavir: Fibrosis: number analyzed (Participants) | 64 | 72 | 71
  Metavir: Fibrosis | 0.02 (0.604) | 0.04 (0.777) | 0.13 (0.653)

15. Secondary Outcome: Mean Change From Baseline in Serum FibroSure (FibroTest/ActiTest) Score at Week 52
Description: FibroTest was for the assessment of fibrosis. Fibro test was calculated using an original combination of five highly concentrated serum biochemical markers; alpha-2-macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin and gammaglutamyltransferase. FibroTest scores range from 0.00 to 1.00 where 0.0-0.21 is no fibrosis and >= 0.59 is cirrhosis. Acti-test was calculated using 6 serum biochemical markers; alpha2macroglobulin, haptoglobin, apolipoprotein A1, total bilirubin, GGT and alanine aminotransferase. ActiTest was used for the assessment of necroinflammatory activity. Test score ranges from 0.00 to 1.00, where 0.00-0.17 indicates no necrosis and >= 0.61 indicates severe necrosis. Day 1 value was considered to be as Baseline value. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing.
Time Frame: Baseline and Week 52
Population: MITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 81 | 80 | 78
Scores on a scale
  FibroSure: Fibrosis Score | -0.004 (0.2187) | -0.064 (0.3032) | -0.103 (0.3044)
  FibroSure: Activity Score | -0.010 (0.1669) | -0.069 (0.2899) | -0.132 (0.2855)

16. Secondary Outcome: Mean Change From Baseline in Serum ALT Levels
Description: ALT was assessed as per upper limit of normal where the normal range was 0-48 international units per liter. Day 1 (before dosing) value was considered to be as Baseline value. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing.
Time Frame: Baseline and Week 52
Population: MITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Per upper limit normal
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 83 | 83 | 80
Per upper limit normal | 0.085 (0.8028) | -0.031 (0.6004) | -0.377 (1.0743)

17. Secondary Outcome: Mean Change From Baseline in Measures of Insulin Resistance
Description: Insulin resistance was measured using Homeostasis Model Assessment of Insulin Resistance (HOMA-IR), Belfiore Insulin Sensitivity Index (ISI) and Quantitative Insulin Sensitivity Check Index (QUICKI). HOMA-IR = fasting plasma insulin*fasting plasma glucose / 22.5 and ISI = 2 / [(fasting plasma glucose from the participant / fasting plasma glucose normal reference range)*( fasting plasma insulin from the participant / fasting plasma insulin normal reference range) + 1] and QUICKI = 1/(log[fasting plasma Insulin] + log[fasting plasma glucose]). Day 1 (before dosing) value was considered to be as Baseline value. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing.
Time Frame: Baseline and Week 52
Population: As Treated Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 60 | 65 | 64
Units on a scale
  HOMA-IR | 0.9743 (6.28858) | -1.3027 (4.73127) | -1.8585 (3.95012)
  QUICKI | -0.0022 (0.01139) | 0.0029 (0.01311) | 0.0070 (0.01106)
  ISI | -0.0451 (0.24469) | 0.0718 (0.28736) | 0.1601 (0.24878)

18. Secondary Outcome: Median Change From Baseline in Serum ALT Over Time
Description: as for outcome 16
Time Frame: Baseline and up to 4 weeks post-treatment (52 weeks)
Population: MITT Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Per upper limit normal
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 88 | 89 | 88
Per upper limit normal
  Week 2: number analyzed (Participants) | 83 | 85 | 84
  Week 2 | -0.021 [-1.063 to 0.833] | -0.083 [-1.688 to 0.854] | -0.167 [-3.458 to 1.458]
  Week 4: number analyzed (Participants) | 83 | 88 | 81
  Week 4 | -0.042 [-1.792 to 1.625] | -0.063 [-2.125 to 0.917] | -0.167 [-5.292 to 1.646]
  Week 10: number analyzed (Participants) | 83 | 87 | 82
  Week 10 | -0.021 [-1.000 to 1.250] | -0.063 [-1.271 to 1.771] | -0.219 [-4.625 to 3.625]
  Week 16: number analyzed (Participants) | 77 | 83 | 81
  Week 16 | 0.021 [-1.417 to 2.583] | -0.125 [-1.292 to 1.104] | -0.208 [-4.000 to 0.917]
  Week 22: number analyzed (Participants) | 76 | 79 | 80
  Week 22 | 0.010 [-1.313 to 2.021] | -0.146 [-1.521 to 1.813] | -0.198 [-5.979 to 1.354]
  Week 28: number analyzed (Participants) | 75 | 78 | 81
  Week 28 | -0.021 [-2.104 to 3.854] | -0.146 [-1.938 to 2.521] | -0.208 [-5.771 to 2.563]
  Week 34: number analyzed (Participants) | 75 | 76 | 78
  Week 34 | -0.042 [-1.313 to 2.979] | -0.188 [-1.854 to 1.583] | -0.271 [-6.188 to 4.042]
  Week 40: number analyzed (Participants) | 72 | 74 | 73
  Week 40 | -0.021 [-1.771 to 4.625] | -0.104 [-2.292 to 1.625] | -0.208 [-3.792 to 2.000]
  Week 46: number analyzed (Participants) | 74 | 71 | 79
  Week 46 | -0.063 [-1.771 to 7.938] | -0.146 [-2.104 to 2.146] | -0.229 [-2.833 to 1.625]
  Week 52: number analyzed (Participants) | 83 | 83 | 80
  Week 52 | 0.021 [-1.917 to 3.542] | -0.083 [-1.396 to 2.021] | -0.271 [-4.125 to 4.042]
  Post-treatment: number analyzed (Participants) | 78 | 73 | 81
  Post-treatment | -0.042 [-2.917 to 6.458] | -0.146 [-2.750 to 1.667] | -0.229 [-3.750 to 4.313]

19. Secondary Outcome: Mean Change From Baseline in Serum Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels at Week 52
Description: Value at Day 1 visit (day of first dose) was considered as Baseline. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing.
Time Frame: Baseline and Week 52
Population: MITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 International unit per milliliter
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 82 | 78 | 82
Log10 International unit per milliliter | -0.020 (0.4264) | -0.006 (0.3760) | 0.040 (0.4803)

20. Secondary Outcome: Median Change From Baseline in Serum HCV RNA Levels Over Time
Description: Serum for HCV RNA levels were collected at pre-screen, Baseline, Week 28, Week 52, and at the 4 week follow up visit. Value at Day 1 visit (day of first dose) was considered as Baseline. Change from Baseline was calculated as the post Baseline assessment minus the Baseline assessment for a given parameter. If either the Baseline or on-treatment value was missing, the change from Baseline value was also set to missing.
Time Frame: Baseline and up to 4 weeks post-treatment (52 weeks)
Population: MITT Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Log10 International unit per milliliter
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
Number analyzed (Participants) | 88 | 89 | 88
Log10 International unit per milliliter
  Week 28: number analyzed (Participants) | 71 | 79 | 79
  Week 28 | 0.112 [-1.02 to 0.82] | 0.011 [-0.93 to 1.61] | 0.071 [-0.62 to 2.41]
  Week 52: number analyzed (Participants) | 82 | 78 | 82
  Week 52 | -0.059 [-0.94 to 1.54] | 0.034 [-0.90 to 1.47] | 0.013 [-0.82 to 2.48]
  Post-treatment: number analyzed (Participants) | 76 | 68 | 78
  Post-treatment | 0.024 [-0.93 to 1.41] | 0.039 [-0.84 to 1.18] | 0.026 [-2.56 to 1.86]

21. Secondary Outcome: Area Under the Plasma Concentration-time Curve During One Dosing Interval of Length 'Tau' (AUC [0-tau]) of GI262570 on Week 2
Description: Samples for Week 2 serial group were collected at 0 (pre-morning dose)1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose. Initially the doses selected for the study were 0.5 mg twice daily and 1.0 mg twice daily. However, because of implementation of Amendment 4, the dose regimen was reduced to half the original dosing resulting in dose once daily.
Time Frame: At 0 (pre-morning dose)1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose on Week 2
Population: The Pharmacokinetic (PK) Parameter Population included all participants in the subset having the serial PK profiles performed at Week 2 and having sufficient data for the calculation of the PK parameters. Initially the doses selected were twice daily, but after implementation of Amendment 4 the dose regimen was reduced to half the original dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanograms per milliliter
Groups:
- GI262570 0.5 mg Twice Daily: Participants in this arm received GI262570 0.5 mg tablet twice daily as per protocol amendment 3. After implementation of protocol 4, they started receiving it once daily. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
- GI262570 0.5 mg Once Daily: Participants received GI262570 0.5 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
- GI262570 1.0 mg Twice Daily: Participants in this arm received GI262570 1.0 mg tablet twice daily as per protocol amendment 3. After implementation of protocol 4, they started receiving it once daily. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
- GI262570 1.0 mg Once Daily: Participants received GI262570 1.0 mg tablet once daily approximately 30 minutes prior to breakfast for 52 weeks. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 8 | 19 | 8 | 14
Hour nanograms per milliliter | 68.65 (64) | 88.87 (34) | 151.11 (55) | 141.03 (29)

22. Secondary Outcome: Dose Normalized (DN) AUC (0-tau) of GI262570 on Week 2
Description: Sample s for Week 2 serial group were collected at 0 (pre-morning dose )1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose. Initially the doses selected for the study were 0.5 mg twice daily and 1.0 mg twice daily. However, because of implementation of Amendment 4, the dose regimen was reduced to half the original dosing resulting in dose once daily.
Time Frame: At 0 (pre-morning dose )1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose on Week 2
Population: PK parameter Population. Initially the doses selected were twice daily, but after implementation of Amendment 4 the dose regimen was reduced to half the original dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours nanograms per milliliter per mg
Groups:
- GI262570 0.5 mg Twice Daily: Participants in this arm received GI262570 0.5 mg tablet twice daily as per protocol amendment 3. After implementation of protocol 4, they started it receiving once daily. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
- GI262570 1.0 mg Twice Daily: Participants in this arm received GI262570 1.0 mg tablet twice daily as per protocol amendment 3. After implementation of protocol 4, they started it receiving once daily. Participant received their morning dose at the site on Weeks 2, 16, 28, 40, and 52.
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 8 | 19 | 8 | 14
Hours nanograms per milliliter per mg | 68.65 (64) | 88.87 (34) | 75.55 (55) | 70.52 (29)

23. Secondary Outcome: Apparent Clearance Following Oral Dosing (CL/F) of GI262570 on Week 2
Description: as for outcome 21
Time Frame: At 0 (pre-morning dose)1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose on Week 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 8 | 19 | 8 | 14
milliliter per hour | 7283.04 (64) | 5626.48 (34) | 6617.76 (55) | 7090.62 (29)

24. Secondary Outcome: Maximum Observed Concentration (Cmax), Minimum Observed Concentration (Cmin) of GI262570 on Week 2
Description: as for outcome 21
Time Frame: At 0 (pre-morning dose)1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose on Week 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 8 | 19 | 8 | 14
Nanograms per milliliter
  Cmax | 21.10 (61) | 30.30 (28) | 49.60 (47) | 50.38 (26)
  Cmin | 0.69 (139) | 0.19 (72) | 1.54 (86) | 0.18 (65)

25. Secondary Outcome: DN Cmax of GI262570 on Week 2
Description: Samples for Week 2 serial group were collected at 0 (pre-morning dose) 1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose. Initially the doses selected for the study were 0.5 mg twice daily and 1.0 mg twice daily. However, because of implementation of Amendment 4, the dose regimen was reduced to half the original dosing resulting in dose once daily.
Time Frame: At 0 (pre-morning dose) 1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose on Week 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter per mg
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 8 | 19 | 8 | 14
Nanograms per milliliter per mg | 21.10 (61) | 30.30 (28) | 24.80 (47) | 25.19 (26)

26. Secondary Outcome: Terminal Elimination Half-life (T1/2), Time to First Quantifiable Concentration (Tlag) and Time to Cmax (Tmax) of GI262570 on Week 2
Description: as for outcome 21
Time Frame: At 0 (pre-morning dose)1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose on Week 2
Population: as for outcome 22
Measure: Median (Full Range); unit: hour
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 8 | 19 | 8 | 14
hour
  T1/2 | 3.33 [1.9 to 4.7] | 2.47 [1.2 to 5.7] | 2.54 [1.6 to 4.4] | 2.25 [1.5 to 4.4]
  Tlag | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  Tmax | 2.00 [1.0 to 6.0] | 1.50 [0.8 to 4.0] | 1.75 [1.0 to 3.9] | 1.75 [0.8 to 4.0]

27. Secondary Outcome: Volume of Distribution Expressed as a Function of Bioavailability (V/F) of GI262570
Description: as for outcome 21
Time Frame: At 0 (pre-morning dose)1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose on Week 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 8 | 19 | 8 | 14
milliliter | 33440.98 (83) | 19971.49 (51) | 25616.42 (85) | 24355.48 (52)

28. Secondary Outcome: GI262570 Serum Concentrations on Week 2, 16, 28, 40, and Week 52
Description: Samples for Week 2 serial group were planned to be collected at 0 (pre-morning dose)1, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 hour post-morning dose. For Weeks 16 and 40 samples were planned to be collected at 0 (pre-morning dose)1 and between 1.5-6 hour post-morning dose 2. For Weeks 28 and 52 samples were planned to be collected at 0 (pre-morning dose)1 and between 6-10 hour post-morning dose 2.
Time Frame: Weeks 2, 16, 28, 40 and 52
Population: PK parameter Population. Initially the doses selected were twice daily, but after implementation of Amendment 4 the dose regimen was reduced to half the original dosing. Data was not collected for this endpoint.
Arm/Group | GI262570 0.5 mg Twice Daily | GI262570 0.5 mg Once Daily | GI262570 1.0 mg Twice Daily | GI262570 1.0 mg Once Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from start of study medication through treatment phase (52 weeks) and assessed up to 56 weeks (4 weeks follow up). SAEs were collected from pre-screening (within 60 days of first dose up to follow up.
Description: AEs and SAEs were reported for the As treated Population which consisted of all participants for whom no clear evidence was available of failure to take study medication.
Arm/Group | Placebo | GI262570 0.5 mg | GI262570 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/89 | 0/88
Serious Adverse Events (participants affected / at risk) | 7/88 | 10/89 | 6/88
Other Adverse Events (participants affected / at risk) | 58/88 | 50/89 | 55/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=88) | GI262570 0.5 mg (N=89) | GI262570 1.0 mg (N=88)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Haemobilia (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Colitis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=88) | GI262570 0.5 mg (N=89) | GI262570 1.0 mg (N=88)
Diarrhoea (Gastrointestinal disorders) | 3 | 10 | 4
Nausea (Gastrointestinal disorders) | 7 | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5 | 2
Constipation (Gastrointestinal disorders) | 5 | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 2 | 5 | 3
Fatigue (General disorders) | 14 | 15 | 10
Oedema peripheral (General disorders) | 13 | 6 | 9
Weight increased (Investigations) | 13 | 17 | 16
Nasopharyngitis (Infections and infestations) | 3 | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 5
Urinary tract infection (Infections and infestations) | 5 | 2 | 1
Headache (Nervous system disorders) | 8 | 9 | 6
Dizziness (Nervous system disorders) | 2 | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 5
Insomnia (Psychiatric disorders) | 5 | 5 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.